CLINICAL TRIAL: NCT03808259
Title: A Randomized, Participant- and Investigator Blind, Double Dummy, Placebo- and Comparator-controlled, Single Ascending Dose and Parallel-group Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Different Modes of (S) Ketamine Administration in Healthy Participants
Brief Title: A Study to Investigate the Different Modes of (S) Ketamine Administration in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: CR108553; 2018-003435-30 (EudraCT Number); 54135419EDI1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-01-04; First posted 2019-01-17 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1: OTF Sublingual and IV (Experimental): Participants will receive (S)-ketamine oral thin film (OTF) at a dose of 7 milligram (mg) [cohort 1], 14 mg [cohort 2], and 28 mg [cohort 3] via sublingual route or 14 mg (S)-ketamine intravenous (IV) infusion for 40 minutes or matching placebo in 1 of 3 serial cohorts. Dose escalation decisions to further cohorts of Part 1 will be made based on safety and tolerability profile of the preceding lower dose level.
  Interventions: Drug: (S)-ketamine Oral Thin Film; Drug: (S)-ketamine IV Infusion; Drug: Placebo
- Part 2: IV Different Infusion Duration (Experimental): Participants will receive single dose (S)-ketamine less than or equal to (<=)14 mg IV at a different infusion duration or matching placebo at a different infusion duration. The infusion duration and dose will be chosen after completion of Part 1.
  Interventions: Drug: (S)-ketamine IV Infusion; Drug: Placebo

INTERVENTIONS:
Drug: (S)-ketamine Oral Thin Film — (S)-ketamine OTF sublingual formulation at a dose of 7 mg, 14 mg, and 28 mg will be administered in sequential cohorts.
  Other Names: JNJ-54135419
  Arms: Part 1: OTF Sublingual and IV
Drug: (S)-ketamine IV Infusion — (S)-ketamine IV solution will be infused at a dose of less than or equal to 14mg.
  Other Names: Ketanest
Drug: Placebo — Participants will receive matching placebo.

SUMMARY:
The purpose of this study is to determine the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of different modes of (S) ketamine administration in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 20 and 28 kilogram per meter square (kg/m^2), inclusive (BMI=weight/height^2) with a minimum weight of 60 kilogram (kg) and a maximum of 100 kg
* Participant must be healthy based on clinical laboratory tests performed at screening. If the results of the serum chemistry panel, hematology or urinalysis are outside the normal reference ranges, retesting of an abnormal lab value(s) that may lead to exclusion will be allowed once during the screening phase
* Participant must be healthy based on physical and neurological examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) (including QT corrected according to Fridericia's formula [QTcF] less than or equal to [<=] 450 milliseconds [msec] for males and <= 470 msec for females) performed at screening. Abnormalities, which are not considered to be of clinical significance by the Investigator, are acceptable. The presence of left bundle branch block (LBBB), atrioventricular (AV) Block (second degree or higher), or a permanent pacemaker or implantable cardioverter defibrillator (ICD) will lead to exclusion
* Participant must have systolic blood pressure (SBP) and heart rate (HR) within normal limits at screening and at Day -1: supine SBP of at least 90 millimeters of mercury (mmHg) and maximum 150mmHg, supine diastolic blood pressure (DBP) should be above 50mmHg and below 90mmHg and the HR must be between 45 beats per minute (BPM) and 100 BPM. If the results are outside the normal reference ranges above, retesting will be allowed once during the screening phase
* Non-smoker (not smoked for 3 months prior to screening)

Exclusion Criteria:

* Cardiac arrhythmias or other cardiac disease, hematological disease, hypertension, lipid abnormalities, respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, Parkinson's disease, infection, or any other illness that the Investigator considers should exclude the participant
* Positive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies or human immunodeficiency virus (HIV) antibodies at screening visit
* Participant has a history of drug or alcohol use disorder or psychiatric disorder according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-V) criteria within 6 months before screening (for example psychotic, bipolar, major depressive, or anxiety disorder) or positive test result(s) for alcohol and/or drugs of abuse (opiates (including methadone), cocaine, amphetamines, methamphetamines, cannabinoids, barbiturates, ecstasy and benzodiazepines) at screening or admission
* Drinks, on average, more than 8 cups of tea/coffee/cocoa/cola per day
* Clinically significant acute illness within 7 days prior to study drug administration

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-09-04 (Actual); Study Completion 2019-09-04 (Actual)

PRIMARY OUTCOMES:
Part 1: Change from Baseline in Clinician-Administered Dissociative States Scale (CADSS) Total Score | Baseline up to Day 1
  CADSS is an instrument for the measurement of present-state dissociative symptoms and will be administered to assess treatment-emergent dissociative symptoms. CADSS consists of 23 subjective items, divided into 3 components: depersonalization (items 3 to 7, 20, and 23), derealization (items 1, 2, 8 to 13, 16 to 19, and 21) and amnesia (items 14, 15, and 22). The participants responses are coded on a 5-point scale (from 0=not at all to 4=extremely). The total score is sum of the 23 items and range from 0 to 92 - best is 0 and worst is 92.
Part 2: Change from Baseline in CADSS Total Score | Baseline up to Day 1
  CADSS is an instrument for the measurement of present-state dissociative symptoms and will be administered to assess treatment-emergent dissociative symptoms. CADSS consists of 23 subjective items, divided into 3 components: depersonalization (items 3 to 7, 20, and 23), derealization (items 1, 2, 8 to 13, 16 to 19, and 21) and amnesia (items 14, 15, and 22). The participants responses are coded on a 5-point scale (from 0=not at all to 4=extremely). The total score is sum of the 23 items and range from 0 to 92 - best is 0 and worst is 92.
Part 1: Number of Participants with Vital Sign Abnormalities | Up to Day 2
  Number of participants with vital signs (Heart Rate and Blood Pressure) abnormalities will be reported.
Part 2: Number of Participants with Vital Sign Abnormalities | Up to Day 2
  Number of participants with vital signs (Heart Rate and Blood Pressure) abnormalities will be reported.
Plasma Concentrations of (S)-ketamine | Part 1: Predose, 1, 3, 5, 10, 15, 30, 40 min, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hour postdose; Part 2: predose, 15, 30 min, 1, 1.6, 2, 3, 3.5, 4, 6, 8, 10, 12, and 24 hours postdose
  Observed plasma concentrations of (S)-ketamine will be reported.
Plasma Concentrations of Nor(S)-ketamine | Part 1: Predose, 1, 3, 5, 10, 15, 30, 40 min, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hour postdose; Part 2: predose, 15, 30 min, 1, 1.6, 2, 3, 3.5, 4, 6, 8, 10, 12 and 24 hours postdose
  Observed plasma concentrations of Nor(S)-ketamine will be reported.
Part 1: Change from Baseline in Electroencephalogram (EEG) Power | Predose (Baseline) and 2.25 hours postdose
  EEG power spectral activity in the alpha 1, alpha 2, beta 1, beta 2, delta, theta and gamma frequency bands will be estimated for the baseline EEG recording and will be compared to the EEG power spectral activity in the same frequency bands.
Part 2: Change from Baseline in EEG Power | Predose (Baseline) and 3.25 hours postdose
  EEG power spectral activity in the alpha 1, alpha 2, beta 1, beta 2, delta, theta and gamma frequency bands will be estimated for the baseline EEG recording and will be compared to the EEG power spectral activity in the same frequency bands.
Part 1: Change from Baseline in Continuous Paired Associate Learning Test (cPALT) Score | Baseline up to Day 1
  The cPALT will be used to assess whether drug will improve performance of complex cognitive tasks. CPAL assesses Visual episodic memory (associate learning) cognitive domain. In this task, participants must learn a series of associations between a set of difficult to verbalize patterns (amoeba) and locations. In participants, 14 pattern/location associations must be learned. In the presentation phase of the task the pattern appears at the location and the participant is required to acknowledge that they have seen the pattern by touching the location at which it appears. Patterns are presented in random order. In the learning phase of the task, participants must place each of the 14 patterns in their correct locations. They must do this in 10 rounds. The outcome is number of errors made in correctly placing each of the four patterns in their location four times (Lower score = better performance).
Part 2: Change from Baseline in cPALT Score | Baseline up to Day 1
  The cPALT will be used to assess whether drug will improve performance of complex cognitive tasks. CPAL assesses Visual episodic memory (associate learning) cognitive domain. In this task, participants must learn a series of associations between a set of difficult to verbalize patterns (amoeba) and locations. In participants, 14 pattern/location associations must be learned. In the presentation phase of the task the pattern appears at the location and the participant is required to acknowledge that they have seen the pattern by touching the location at which it appears. Patterns are presented in random order. In the learning phase of the task, participants must place each of the 14 patterns in their correct locations. They must do this in 10 rounds. The outcome is number of errors made in correctly placing each of the four patterns in their location four times (Lower score = better performance).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency